CLINICAL TRIAL: NCT01904084
Title: A Randomized, Prospective Comparison of Volar Locked Plating Versus Hoffman II Bridging External Fixation in Patients With Dislocated Distal Radius Fractures, AO/OTA Type A.
Brief Title: Volar Locked Plating vs Bridging External Fixation in Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/555
Record Dates: First submitted 2013-06-20; First posted 2013-07-22 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2017-06

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volar locked plating (Active Comparator): One group with distal radius fracture is operated with Locking plate
  Interventions: Device: Volar locked plating
- Hoffman external fixator (Active Comparator): One group with distal radius fracture is operated with Hoffman external fixator
  Interventions: Device: Hoffman external fixator

INTERVENTIONS:
Device: Volar locked plating — Operative treatment of distal radius fracture with volar locking plate
  Other Names: DVR Anatomic plate, Hand Innovations, De Puy
  Arms: Volar locked plating
Device: Hoffman external fixator — Patients with distal radius fracture operated with Hoffman external fixator
  Other Names: Bridging Hoffman II Compact, Stryker
  Arms: Hoffman external fixator

SUMMARY:
The purpose of this study is to evaluate function, pain and radiographic evaluation in patients treated with volar locked plating versus Hoffman II bridging external fixation in patients with extraarticular distal radius fractures, AO/OTA type A

DETAILED DESCRIPTION:
We have designed a randomized prospective study for comparison of volar locked plating versus Hoffman II bridging external fixation in patients with extraarticular dislocated distal radius fractures AO/OTA type A3. On the basis of power analysis a total of 160 patients are to be included in this project. The follow-up period is 1 year and evaluation is based on x-ray analysis, grip strength, range of motion, pain and satisfaction with the treatment ( PRWE, Quick-DASH)

ELIGIBILITY:
Inclusion Criteria:

* Patients with dislocated extraarticular distal radius fracture age 18-70 years

Exclusion Criteria:

* Cognitively impaired
* Drug abuse
* Congenital bone disease
* Earlier wrist injury
* Open fracture, Gustilo-Anderson type 3
* Pathological fractures( except osteoporotic fractures)
* Tourists

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-08; Primary Completion 2017-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Patient rated wrist evaluation (PRWE)score | 3 months
Patient rated wrist evaluation (PRWE)score | 6 weeks
Patient rated wrist evaluation (PRWE)score | 12 months

SECONDARY OUTCOMES:
Quick-DASH score | 6 weeks, 3 and 12 months
Pain VAS-score | 6 weeks, 3 and 12 months
Complications | 6 weeks, 3 and 12 months
  Number of patients with per- and postoperative complications will be registrated. Types of expected complications: Tendon rupture, Tendon irritation, Carpal Tunnel Syndrome, Complex Regional Pain Syndrome, Screw displacement/screw loosening, Delayed fracture union
Radiographic evaluation | 6 weeks and 12 months
  Palmar tilt, Radial inclination, Ulnar variance, Fracture union

CONTACTS AND LOCATIONS:
Overall Officials: Trine Ludvigsen, Md, Principal Investigator
Locations (1):
- Orthopaedic depatment, Voss hospital, Bergen, Voss, Norway

REFERENCES:
- [Background] Esposito J, Schemitsch EH, Saccone M, Sternheim A, Kuzyk PR. External fixation versus open reduction with plate fixation for distal radius fractures: a meta-analysis of randomised controlled trials. Injury. 2013 Apr;44(4):409-16. doi: 10.1016/j.injury.2012.12.003. Epub 2013 Jan 6. PMID 23298757
- [Derived] Ludvigsen T, Matre K, Vetti N, Kristoffersen PM, Toppe MK, Gudmundsdottir R, Krukhaug Y, Dybvik E, Fevang JM. Is there a correlation between functional results and radiographic findings in patients with distal radius fracture A0 type A3 treated with volar locking plate or external fixator? OTA Int. 2021 Aug 9;4(3):e142. doi: 10.1097/OI9.0000000000000142. eCollection 2021 Sep. PMID 34746674